CLINICAL TRIAL: NCT01457703
Title: Reproductive Hormonal Alterations in Obesity, AIMS #1 & #2
Brief Title: Reproductive Hormonal Alterations in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 09-0977; U54HD058155 (NIH)
Record Dates: First submitted 2011-09-21; First posted 2011-10-24 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: LH pulsatility; Obesity; Reproduction
MeSH Terms: conditions — Obesity | interventions — cetrorelix; Gonadotropin-Releasing Hormone; Luteinizing Hormone, beta Subunit; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMI ≥30 kg/m2 (Active Comparator): Group 2:
  * BMI ≥30 kg/m2
  * History of regular menstrual cycles every 25-40 days
  Gonadorelin-GnRH (Lutrepulse), GnRH antagonists - Cetrorelix (Cetrotide), Recombinant LH (Luveris) were administered in Aim 1. GnRH or gonadorelin (Lutrepulse) and Letrozole were administered in Aim 2.
  Interventions: Drug: Cetrorelix; Drug: Gonadorelin-GnRH; Drug: Recombinant LH; Drug: Letrozole
- BMI 18-25 kg/m2 (Experimental): * BMI 18-25 kg/m2
  * History of regular menstrual cycles every 25-35 days
  Gonadorelin-GnRH (Lutrepulse), GnRH antagonists - Cetrorelix (Cetrotide), Recombinant LH (Luveris) were administered in Aim 1. GnRH or gonadorelin (Lutrepulse) and Letrozole were administered in Aim 2.
  Interventions: Drug: Cetrorelix; Drug: Gonadorelin-GnRH; Drug: Recombinant LH; Drug: Letrozole

INTERVENTIONS:
Drug: Cetrorelix — Abolishes pituitary sensitivity to GnRH.
  Other Names: Cetrotide
Drug: Gonadorelin-GnRH — GnRH is used to stimulate the pituitary gland to produce LH and FSH.
  Other Names: Lutrepulse
Drug: Recombinant LH — Used to stimulate ovarian function in women.
  Other Names: Luveris
Drug: Letrozole — An aromatase inhibitor.
  Other Names: Femara

SUMMARY:
The purpose of this study is to determine why obese women have lower hormone levels and less fertility than women of normal body weight. The proposal will examine the reproductive system at the level of the brain and the ovary to define the changes that happen leading to lowered hormone production. Women will be studied throughout a menstrual cycle and given medications that will test how well their pituitary gland can make hormones that stimulate the ovary (luteinizing hormone (LH) and follicle stimulating hormone (FSH)). They will also be given a medication to abolish estrogen production in the body and their response to this medication will be assessed. Finally, the ovary's ability to produce progesterone after ovulation will be examined.

--Hypotheses:

1. Obese women have reduced pituitary sensitivity to exogenous gonadotropin-releasing hormone (GnRH), but normal clearance of exogenous LH. (comparative study of obese compared to normal weight women)
2. Obese women have abnormally increased sensitivity to estradiol negative feedback which will be reversed by an aromatase inhibitor. (comparative study of obese compared to normal weight women)

DETAILED DESCRIPTION:
AIM 1: test the hypothesis that reduced pituitary sensitivity to GnRH-induced LH and FSH secretion causes the relative hypogonadotropic hypogonadism of obesity AIM 2: test the hypothesis that the hypothalamic-pituitary axis is abnormally sensitive to estradiol negative feedback in obesity

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 at study entry
* BMI either 18-25 kg/m2 or ≥30 kg/m2
* prolactin (PRL) and thyroid-stimulating hormone (TSH) within normal laboratory ranges at screening
* Baseline hemoglobin >11 gm/dl
* History of regular menstrual cycles every 25-35 days if BMI 18-25 kg/m2
* History of regular menstrual cycles every 25-40 days if BMI ≥30 kg/m2

Exclusion Criteria:

* History of chronic disease affecting hormone production, metabolism or clearance
* Use of medications that are known to alter or interact with reproductive hormones (e.g., thiazolidinediones, metformin)
* Use of hormones within three months of enrollment
* Excessive exercise (>4 hours per week)
* Pregnancy, breast-feeding or current active attempts to conceive

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Santoro, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Clinical Translational Research Center, Aurora, Colorado, United States

REFERENCES:
- [Background] Jain A, Polotsky AJ, Rochester D, Berga SL, Loucks T, Zeitlian G, Gibbs K, Polotsky HN, Feng S, Isaac B, Santoro N. Pulsatile luteinizing hormone amplitude and progesterone metabolite excretion are reduced in obese women. J Clin Endocrinol Metab. 2007 Jul;92(7):2468-73. doi: 10.1210/jc.2006-2274. Epub 2007 Apr 17. PMID 17440019
- [Background] Haynes G, Bailey MK, Davis S, Mahaffey JE. Use of methylprednisolone in epidural analgesia. Arch Neurol. 1989 Nov;46(11):1167-8. doi: 10.1001/archneur.1989.00520470017014. No abstract available. PMID 2818247
- [Background] Rochester D, Jain A, Polotsky AJ, Polotsky H, Gibbs K, Isaac B, Zeitlian G, Hickmon C, Feng S, Santoro N. Partial recovery of luteal function after bariatric surgery in obese women. Fertil Steril. 2009 Oct;92(4):1410-1415. doi: 10.1016/j.fertnstert.2008.08.025. Epub 2008 Sep 30. PMID 18829008
- [Background] Santen RJ, Bardin CW. Episodic luteinizing hormone secretion in man. Pulse analysis, clinical interpretation, physiologic mechanisms. J Clin Invest. 1973 Oct;52(10):2617-28. doi: 10.1172/JCI107454. PMID 4729055
- [Derived] Roth LW, Allshouse AA, Lesh J, Polotsky AJ, Santoro N. The correlation between self-reported and measured height, weight, and BMI in reproductive age women. Maturitas. 2013 Oct;76(2):185-8. doi: 10.1016/j.maturitas.2013.07.010. Epub 2013 Aug 16. PMID 23958434
- See also: PI Biographical data — http://www.cudoctors.com/find-a-doctor/profile/?providerID=3067&name=santoro

RESULTS

PARTICIPANT FLOW:
Groups:
- BMI ≥30 kg/m2: * BMI ≥30 kg/m2
  * History of regular menstrual cycles every 25-40 days
  Letrozole, Gonadorelin-GnRH, Luveris-lutropin, cetrorelix: Reproductive Hormonal Alterations in Obesity, Aims #1 and 2" Description: comparative study of pathophysiology
- BMI 18-25 kg/m2: * BMI 18-25 kg/m2
  * History of regular menstrual cycles every 25-35 days
  Letrozole, Gonadorelin-GnRH, Luveris-lutropin, cetrorelix: Reproductive Hormonal Alterations in Obesity, Aims #1 and 2" Description: comparative study of pathophysiology
Period: Overall Study
Arm/Group | BMI ≥30 kg/m2 | BMI 18-25 kg/m2
Started | 29 | 33
Completed | 23 | 22
Not Completed | 6 | 11
Not completed — Screen Failure | 5 | 7
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMI ≥30 kg/m2 | BMI 18-25 kg/m2 | Total
Number analyzed (Participants) | 29 | 33 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 33 | 62
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 24 | 28 | 52
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 15 | 19 | 34
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 29 | 33 | 62

OUTCOME MEASURES:

1. Primary Outcome: Changes in Luteinizing Hormone (LH) Pulse Amplitude (Aim 1)
Description: Luteinizing Hormone (LH) Pulse Amplitude was measured hourly during the 12 hour study visit, and was compared between the obese and normal weight groups.
Time Frame: Measured hourly and averaged over the 12 hour study visit
Population: This study was divided into two aims, and 10 obese and 10 normal weight women completed the study procedures and contributed data for analyses related to Aim 1.
Measure: Mean (Inter-Quartile Range); unit: IU/L
Arm/Group | BMI ≥30 kg/m2 | BMI 18-25 kg/m2
Number analyzed (Participants) | 10 | 10
IU/L | 4.1 [2.9 to 5.2] | 3.6 [2.7 to 9.9]

2. Primary Outcome: Changes in Luteinizing Hormone (LH) Pulse Amplitude (Aim 2)
Description: as for outcome 1
Time Frame: Measured hourly and averaged over the 12 hour study visit
Population: This study was divided into two aims, and only 12 obese and 11 normal weight women completed the study procedures for Aim 2 that allowed measure of LH pulse amplitude.
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- BMI ≥30 kg/m2: * BMI ≥30 kg/m2
  * History of regular menstrual cycles every 25-40 days
  GnRH or gonadorelin (Lutrepulse) and Letrozole were administered in Aim 2. Description: comparative study of pathophysiology
- BMI 18-25 kg/m2: * BMI 18-25 kg/m2
  * History of regular menstrual cycles every 25-35 days
  GnRH or gonadorelin (Lutrepulse) and Letrozole were administered in Aim 2. Description: comparative study of pathophysiology
Arm/Group | BMI ≥30 kg/m2 | BMI 18-25 kg/m2
Number analyzed (Participants) | 12 | 11
IU/L | 2.21 (.32) | 4.44 (1.03)

3. Primary Outcome: Changes in Pregnanediol Glucuronide (PdG) (Aim 2)
Description: Pregnanediol glucuronide (PdG) was collected daily over the course of one menstrual cycle and averaged.
Time Frame: Averaged over the length of menstrual cycle
Population: This study was divided into two aims, and only 12 obese and 10 normal weight women completed the urine collection study procedures for Aim 2 that allowed measure of PdG.
Measure: Mean (Standard Deviation); unit: ug/cycle
Arm/Group | BMI ≥30 kg/m2 | BMI 18-25 kg/m2
Number analyzed (Participants) | 12 | 10
ug/cycle | 54.1 (33) | 88.7 (64.6)

4. Secondary Outcome: Changes in Follicle Stimulating Hormone (FSH) (Aim 1)
Description: Follicle-stimulating hormone was measured hourly during the 12 hour study visit, and was compared between the obese and normal weight groups.
Time Frame: Measured hourly and averaged over the 12 hour study visit
Population: This study was divided into two aims, and only 10 obese and 10 normal weight women completed the study procedures for Aim 1 that allowed measure of FSH.
Measure: Mean (Inter-Quartile Range); unit: IU/L
Arm/Group | BMI ≥30 kg/m2 | BMI 18-25 kg/m2
Number analyzed (Participants) | 10 | 10
IU/L | 3.8 [2.1 to 4.2] | 3.3 [3 to 4.9]

5. Secondary Outcome: Changes in Follicle Stimulating Hormone (FSH) (Aim 2)
Description: as for outcome 4
Time Frame: Measured hourly and averaged over the 12 hour study visit
Population: This study was divided into two aims, and only 12 obese and 11 normal weight women completed the study procedures for Aim 2 that allowed measure of FSH.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | BMI ≥30 kg/m2 | BMI 18-25 kg/m2
Number analyzed (Participants) | 12 | 11
IU/L | 5.31 (.38) | 6.18 (.94)

ADVERSE EVENTS:
Arm/Group | BMI ≥30 kg/m2 | BMI 18-25 kg/m2
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/33
Other Adverse Events (participants affected / at risk) | 0/29 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No